CLINICAL TRIAL: NCT01025024
Title: Investigation of Genetic Disease Marker Associated With Korean Glaucoma Patients Patients, A Single-nucleotide Polymorphism(SNP)Analysis for Primary Open Angle Glaucoma
Brief Title: Investigation of Genetic Disease Marker Associated With Korean Glaucoma Patients
Status: Completed | Type: Observational
Sponsor: Chungnam National University (Other)
Collaborators: Korea Healthcare Technology R&D Project (Unknown); Korea Advanced Institute of Science and Technology (Other)
Responsible Party: Chang-sik Kim, professor, Department of Ophthalmology, College of Medicine, Chungnam National University
Other Study IDs: CNUH81510-886; A080587 (Other Grant/Funding Number: Korea Healthcare Technology R&D Project)
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Single-nucleotide Polymorphism (SNP) for Glaucoma
Keywords: SNP; single-nucleotide polymorphism; glaucoma; primary open angle glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- POAG group: Elevated intraocular pressure normal open angle glaucomatous optic nerve head abnormality glaucomatous visual field defect
  Interventions: Genetic: SNP analysis of the DNA
- Normal control: Normal intraocular pressure No optic disc abnormality No visual field defect No significant ocular and systemic disease
  Interventions: Genetic: SNP analysis of the DNA

INTERVENTIONS:
Genetic: SNP analysis of the DNA — SNP analysis of the DNA obtained from peripheral blood sample

SUMMARY:
A single-nucleotide polymorphism (SNP) analysis of DNA obtained from peripheral blood of the glaucoma patients and the normal control will be performed to find genetic marker for primary open angle glaucoma.

DETAILED DESCRIPTION:
Unrelated Korean subjects who have primary open angle glaucoma were recruited in the current study. Genotyping for various SNP associated with POAG due to the linkage disequilibrium patterns is to be performed. Genotypes would be statistically compared between patients with primary open angle glaucoma and normal control subjects free of any eye diseases.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary open angle glaucoma

Exclusion Criteria:

* Primary open angle glaucoma combined with congenital ocular disease
* Primary open angel glaucoma combined with other ocular disease
* Significant systemic disease other than systemic hypertension and diabetes

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with open angle glaucoma who visited glaocoma clinic of departemtn of Ophtalmology, Chungnam National University Hospital, Daejeon, south Korea
Sampling Method: Non-Probability Sample
Enrollment: 1224 (Actual)
Dates: Start 2007-01; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
genotyping for the SNP associated with primary open angle glaucoma | one year

SECONDARY OUTCOMES:
genotyping for rs7961953 and additional SNPs in TMTC2 from other linkage disequilibrium patterns | one year

CONTACTS AND LOCATIONS:
Overall Officials: Chang-sik Kim, professor, Principal Investigator — Department of Ophthalmology, Chungnam National University Hospital; Changwon Kang, professor, Study Chair — Korea Advanced Institute of Science and Technology; Kyunglan Kim, Study Director — Department of Biological Sciences, Korea Advanced Institute of Science and Technology
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea